CLINICAL TRIAL: NCT05218551
Title: Comparison of Different Objective Nociceptive Measurement Methods During General Anesthesia or Sedation Under Surgery
Brief Title: Comparison of Different Objective Nociceptive Measurement Methods During Surgery
Status: Completed | Type: Observational
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-03692
Record Dates: First submitted 2022-01-15; First posted 2022-02-01 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Nociceptive Pain
MeSH Terms: conditions — Nociceptive Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Traditionally, hemodynamic response e.g. pulse and blood pressure are used to evaluate pain in humans who are anesthetized. These values, however, can be affected by factors other than pain response . In this observational study, different types of digital methods are used that can distinguish signs of pain. However, the study aim to collect data and correlate in between different methods to ensure its reliability.

DETAILED DESCRIPTION:
In humans who undergoing anesthesia or only receiving sedation with the addition of painkillers medication under surgery. Nociceptive response usually treats on the basis of hemodynamic and/or respiratory changes. These are interpreted together with a number of other parameters. The anesthetist can't be totally sure if it is nociceptive response or to light anesthesia given. Today, there are new monitors included techniques for measuring pain (nociception), but these are not used routinely.

By put sensors (adhesive patches) on the skin and connect to these new devices perhaps the anesthetist can be more sure what stimuli patient are responding from, pain or light anesthesia.

These techniques measure muscle activity including sweat gland which have been shown in other research studies demonstrate a higher accuracy regarding the response to nociception. The parameters are presented on a monitor as a value, 0-10 or 0-100. This research study is an observational study and intends to observe values / figures that arise from two different types of commercial monitors and manufactures. After the anesthesia, these values will be compared and evaluated in resect as well to hemodynamic response and in between monitors. The two techniques have never before been studied simultaneously on the same human been (control).

ELIGIBILITY:
Inclusion Criteria:

* All patients over 18 yrs old,
* Patients who will be anesthetized or sedated under intervention surgery or surgery

Exclusion Criteria:

* Not speaking Swedish
* Neuro cognitive diorders e.g. dementia or can't respond on information given.
* Chronic pain
* Acute brain trauma
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ° Patients over 18 yrs old, who will be anesthetized or sedated under intervention surgery or surgery.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2022-01-02 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
An index will be observed 0-100 and hemodynamic response, heart rate and blood pressure. | numbers will be collected every minute during the surgery often 1 hour
  Data collect only numbers. These are going to be correlated.

CONTACTS AND LOCATIONS:
Overall Officials: Pether Jildenstål, Prof., Study Director — Göteborg University
Locations (1):
- Sahlgrenska University hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Norbeck DW, Lindgren S, Wolf A, Jildenstal P. Reliability of nociceptive monitors vs. standard practice during general anesthesia: a prospective observational study. BMC Anesthesiol. 2025 Jan 31;25(1):51. doi: 10.1186/s12871-025-02923-4. PMID 39891061